CLINICAL TRIAL: NCT02744196
Title: Multicenter Comparative Randomised Double-blind Placebo-controlled Clinical Trial to Evaluate Efficacy and Safety of Acellbia® (JSC "BIOCAD") With Methotrexate in First Line of Biological Therapy of Patients With Active Rheumatoid Arthritis
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of Acellbia® (JSC "BIOCAD") With Methotrexate in First Line Biological Therapy of Patients With Active Rheumatoid Arthritis
Acronym: ALTERRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-020-4
Record Dates: First submitted 2016-04-04; First posted 2016-04-20 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; rheumatism; Acellbia; methotrexate; biologic therapy; monoclonal antibody; rituximab
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases | interventions — Rituximab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acellbia + methotrexate (Experimental): 106 patients of this group will receive methotrexate in combination with a drug Acellbia to be used at a dose of 600 mg as a slow intravenous infusion carried out on day 1 and day 15.
  If a follow-up examination at 24 weeks or later (up to 48 weeks) reveals that the patient still has active arthritis (evaluation index DAS28-4 (ESR)> 2,6 points), the therapy with Acellbia is repeated by the same scheme - 2 infusion at a dose of 600 mg at intervals of 14 days.
  Interventions: Biological: Acellbia; Drug: Methotrexate
- Placebo + methotrexate (Placebo Comparator): 53 patients of this group will receive methotrexate in combination with a placebo to be used as a slow intravenous infusion carried out on day 1 and day 15.
  If a follow-up examination at 24 weeks or later (up to 48 weeks) reveals that the patient still has active arthritis (evaluation index DAS28-4 (ESR)> 2,6 points), the patient receives open therapy with Acellbia is initiated: 2 infusion at a dose of 600 mg at intervals of 14 days.
  Interventions: Biological: Acellbia; Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Biological: Acellbia — Acellbia is rituximab biosimilar, monoclonal antibody which binds CD20.
  Other Names: rituximab
Drug: Placebo — Placebo solution will look identical to the Acellbia solution.
  Arms: Placebo + methotrexate
Drug: Methotrexate

SUMMARY:
The mail goal of this study is to establish superiority in efficacy of Acellbia® applied in a dose of 600 mg (Day 1 and Day 15) in combination with methotrexate in patients with active RA seropositive previously untreated with biological therapy, compared to standard therapy with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent. Age from 18 to 80 years. Rheumatoid arthritis diagnosed at least 6 months before informed consent signing Presence of more than 8 swollen and more than 8 painful joints at screening. C-reactive protein 7 mg/l or more AND/OR erythrocyte sedimentation rate 28 mm/hour or more.

Antibodies to citrullinated cyclic peptide 20 U/ml or more AND/OR rheumatoid factor-IgM higher than upper normal limit.

Documented regular methotrexate intake for 12 weeks, stable dose from 10 to 25 mg/week during last 4 weeks before signing informed consent.

Exclusion Criteria:

Methotrexate intolerance. Felty's syndrome. Patient functional status - IV class according to ACR. Previous use of biologic drugs to treat rheumatoid arthritis, biologic drugs that deplete CD20-lymphocytes, azathioprine use in the last 28 days prior to informed consent signing, leflunomide use in the last 8 weeks prior to informed consent signing, sulphasalazine/hydroxyquinoline use in the last 28 days prior to informed consent signing, intraarticular use of corticosteroids in the last 4 weeks prior to informed consent signing, patient requires prednisolone (or analogues) in a dose more than 10 mg/day or dose is unstable during 4 weeks prior to informed consent signing, requirement in non-steroid antiinflammatory drugs if their dose was not stable during last 8 weeks prior to informed consent signing.

Patient has inflammatory joint disease otherwise than rheumatoid arthritis or systemic autoimmune diseases.

Full list of inclusion and exclusion criteria can be found in Study Protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who developed ACR20 response on 24 week of therapy | Week 24
  The proportion of patients achieving at least a 20% improvement in ACR criteria at 24 weeks of therapy.

SECONDARY OUTCOMES:
Percentage of patients who developed ACR50 and ACR70 response on 24 week of therapy | Week 24
  The proportion of patients achieving at least 50% and 70% improvement in ACR criteria at 24 weeks of therapy.
Percentage of patients who developed ACR20, ACR50 and ACR70 response on 16 week of therapy | Week 16
  The proportion of patients achieving at least 20%, 50% and 70% improvement in ACR criteria after 16 weeks of therapy.
Change in average DAS28-4 (ESR) score after 24 weeks of therapy | Week 24
  Change in average DAS28-4 (ESR) score after 24 weeks of therapy
Change in average HAQ-DI score after 24 weeks of therapy | Week 24
Change in average score according to modified Sharp method of assessment after 24 weeks of therapy | Week 24
Change in average score of erosions according to modified Sharp method of assessment after 24 weeks of therapy | Week 24
Change in average score of joint spase narrowing according to modified Sharp method of assessment after 24 weeks of therapy | Week 24
Percentage of patients with progression of disease according to modified Steinbrocker method of assessment after 24 weeks of treatment | Week 24
Percentage of patients who developed ACR20, ACR50 and ACR70 response on 52 week of therapy | Week 52
  The proportion of patients achieving at least 20%, 50% and 70% improvement in ACR criteria after 52 weeks of therapy.
Change in average DAS28-4 (ESR) score after 52 weeks of therapy | Week 52
  Change in average DAS28-4 (ESR) score after 52 weeks of therapy
Change in average HAQ-DI score after 52 weeks of therapy | Week 52
Change in average score according to modified Sharp method of assessment after 52 weeks of therapy | Week 52
Change in average score of erosions according to modified Sharp method of assessment after 52 weeks of therapy | Week 52
Change in average score of joint space narrowing according to modified Sharp method of assessment after 52 weeks of therapy | Week 52
Percentage of patients with progression of disease according to modified Steinbrocker method of assessment after 52 weeks of treatment | Week 52
Frequency and severity of AE/SAE | 52 weeks
  Frequency and severity of AE/SAE in patients who received at least one injection of study drug/placebo
Frequency of AE 3-4 grade CTCAE 4.03 | 52 weeks
  Frequency of AE 3-4 grade CTCAE 4.03 in patients who received at least one injection of study drug/placebo
Frequency of premature withdrawal due to AE/SAE | 52 weeks
Percentage of patients who have developed binding and neutralizing antibodies to rituximab on week 24 and week 52 | Week 24, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD

IPD SHARING:
Plan to Share IPD: Undecided